CLINICAL TRIAL: NCT02352090
Title: Synthetic vs Natural Estrogen in Combined Oral Contraception- Effect on Insulin Sensitivity, Coagulation, Inflammation and Endometrium - a Comparison With a Progestin-only Preparation.
Brief Title: Synthetic vs Natural Estrogen in Combined Oral Contraception
Acronym: SYLVI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Annina Haverinen, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SYLVI030785
Record Dates: First submitted 2015-01-20; First posted 2015-02-02 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Contraception
Keywords: Contraception, oral; Ethinyl Estradiol; Estradiol Valerate; Dienogest; Insulin resistance; Chronic inflammation; Coagulation
MeSH Terms: conditions — Insulin Resistance; Thrombosis | interventions — Ethinyl Estradiol; dienogest; estradiol valerate-dienogest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Synthetic estrogen + progestin (Experimental): Ethinyl estradiol / dienogest
  Interventions: Drug: Ethinyl estradiol / dienogest
- Natural estrogen + progestin (Experimental): Estradiol valerate / dienogest
  Interventions: Drug: Estradiol valerate / dienogest
- Progestin-Only (Active Comparator): Dienogest
  Interventions: Drug: Dienogest

INTERVENTIONS:
Drug: Ethinyl estradiol / dienogest — One tablet orally for 9 weeks, continuous use
  Other Names: Valette, ATC code G03AA
  Arms: Synthetic estrogen + progestin
Drug: Estradiol valerate / dienogest — One tablet orally for 9 weeks, continuous use
  Other Names: Qlaira, ATC code G03AB08
  Arms: Natural estrogen + progestin
Drug: Dienogest — One tablet orally for 9 weeks, continuous use
  Other Names: Visanne, ATC code G03D
  Arms: Progestin-Only

SUMMARY:
The main objective of the study is to compare the metabolic effects of natural estradiol and synthetic ethinylestradiol used in combined oral contraception in healthy women. A progestin-only preparation will be used in comparison. The main goal is to study the effects on glucose metabolism, coagulation and a markers of chronic inflammation (such as hs-CRP). Our hypothesis is that the natural estradiol preparation will influence blood glucose levels, markers of coagulation and chronic inflammation less than the ethinylestradiol preparation. The progestin-only preparation will not effect these parameters.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-24.9, regular menstrual cycles (21-35 days), a minimum of 2 months without any hormonal contraceptives, no contraindications for use of hormonal contraception

Exclusion Criteria:

* Polycystic ovaries, hypertension, smoking, alcohol abuse, pregnancy, lactation, abnormal result in pre-screening 2h oral glucose tolerance test, regular medications

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oskari Heikinheimo, Prof., PhD., MD., Study Chair — Helsinki University Central Hospital, Department of Gynecology and Obstetrics. Helsinki Univeristy, Medical Faculty; Juha Tapanainen, Prof., PhD, MD., Study Chair — Helsinki University Central Hospital, Department of Gynecology and Obstetrics. Helsinki Univeristy, Medical Faculty; Terhi Piltonen, PhD, MD, Principal Investigator — Oulu University Hospital, Department of Gynecology and Obstetrics; Annina Haverinen, MD, PhD student, Principal Investigator — Helsinki University Central Hospital, Department of Gynecology and Obstetrics. Helsinki University, Faculty of Medicine
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Kätilöopisto Maternity Hospital, Helsinki
  - Oulu University Hospital, Department of Gynecology and Obstetrics, Oulu

REFERENCES:
- [Derived] Kangasniemi MH, Arffman RK, Joenvaara S, Haverinen A, Luiro K, Tohmola T, Renkonen R, Heikinheimo O, Tapanainen JS, Piltonen TT. Ethinylestradiol in combined hormonal contraceptive has a broader effect on serum proteome compared with estradiol valerate: a randomized controlled trial. Hum Reprod. 2023 Jan 5;38(1):89-102. doi: 10.1093/humrep/deac250. PMID 36416543
- [Derived] Kangasniemi MH, Arffman RK, Haverinen A, Luiro K, Hustad S, Heikinheimo O, Tapanainen JS, Piltonen TT. Effects of estradiol- and ethinylestradiol-based contraceptives on adrenal steroids: A randomized trial. Contraception. 2022 Dec;116:59-65. doi: 10.1016/j.contraception.2022.08.009. Epub 2022 Sep 7. PMID 36084710
- [Derived] Haverinen AH, Luiro KM, Szanto T, Kangasniemi MH, Hiltunen L, Sainio S, Piltonen TT, Lassila R, Tapanainen JS, Heikinheimo O. Combined oral contraceptives containing estradiol valerate vs ethinylestradiol on coagulation: A randomized clinical trial. Acta Obstet Gynecol Scand. 2022 Oct;101(10):1102-1111. doi: 10.1111/aogs.14428. Epub 2022 Jul 31. PMID 35909329
- [Derived] Kangasniemi MH, Haverinen A, Luiro K, Hiltunen JK, Komsi EK, Arffman RK, Heikinheimo O, Tapanainen JS, Piltonen TT. Estradiol Valerate in COC Has More Favorable Inflammatory Profile Than Synthetic Ethinyl Estradiol: A Randomized Trial. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa186. doi: 10.1210/clinem/dgaa186. PMID 32303765

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Started | 20 | 20 | 19
Completed | 19 | 20 | 17
Not Completed | 1 | 0 | 2
Not completed — general malaise | 1 | 0 | 0
Not completed — non-specified mild side-effects | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only | Total
Number analyzed (Participants) | 19 | 20 | 17 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (3.8) | 24.1 (3.6) | 24.0 (3.9) | 24.6 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 17 | 56
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 20 | 17 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 63.3 (4.5) | 61.4 (5.8) | 58.0 (7.1) | 61.0 (6.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (1.9) | 22.4 (1.6) | 21.9 (1.9) | 22.5 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Matsuda Index- Whole Body Insulin Sensitivity Index
Description: Matsuda index is calculated from the standard 2h Oral Glucose Tolerance Test and corresponding insulin values.
  Matsuda index = 10,000/square root of [fasting glucose x fasting insulin] x [mean glucose x mean insulin during OGTT]) The Matsuda index is correlated (r = 0.73) with the rate of whole-body glucose disposal during the euglycemic insulin clamp.
  Matsuda index <2.5 is considered insulin resistant, higher values indicate less insulin resistance. A decrease in matsuda index over the study period would indicate decreased insulin sensitivity.
Time Frame: We calculated the change in Matsuda index from baseline to 9 weeks.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 19 | 20 | 17
units on a scale | -1.02 [-2.51 to 0.46] | -0.10 [-1.34 to 1.14] | -1.45 [-3.22 to 0.32]
Statistical Analysis 1: Comparison: Synthetic Estrogen + Progestin vs Natural Estrogen + Progestin vs Progestin-Only; Test type: Other; p = 0.27, ANOVA

2. Secondary Outcome: Fasting Insulin
Description: Mean change in fasting serum insulin from baseline to nine weeks
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: mU/l
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 19 | 20 | 17
mU/l | 1.4 [-0.45 to 3.24] | 1.02 [-0.6 to 2.6] | 1.99 [0.33 to 3.65]

3. Secondary Outcome: High-sensitivity C Reactive Protein
Description: Change in plasma concentrations of acute phase protein 'C reactive protein' (CRP), a marker of chronic inflammation.
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 19 | 20 | 17
mg/L | 1.10 [0.05 to 2.15] | -0.06 [-0.54 to 0.42] | 0.13 [-0.22 to 0.48]

4. Secondary Outcome: Total Cholesterol
Description: Change in concentrations of total cholesterol from baseline to nine weeks
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 19 | 20 | 17
mmol/L | 0.10 [-0.18 to 0.38] | -0.16 [-0.33 to 0.02] | 0.11 [-0.11 to 0.32]

5. Secondary Outcome: Low-Density Lipoprotein (LDL)
Description: Change in concentration of Low-Density Lipoprotein LDL from baseline to nine weeks
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 19 | 20 | 17
mmol/L | -0.16 [-0.41 to 0.08] | -0.14 [-0.31 to 0.04] | 0.01 [-0.19 to 0.21]

6. Secondary Outcome: High-Density Lipoprotein (HDL)
Description: Change in concentration of High-Density Lipoprotein HDL from baseline to nine weeks
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 19 | 20 | 17
mmol/L | 0.20 [0.09 to 0.31] | -0.02 [-0.11 to 0.07] | -0.02 [-0.11 to 0.07]

7. Secondary Outcome: Triglyceride
Description: Change in triglyceride concentrations from baseline to nine weeks
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 19 | 20 | 17
mmol/L | 0.45 [0.35 to 0.56] | 0.18 [0.01 to 0.35] | 0.06 [-0.04 to 0.15]

8. Secondary Outcome: D-dimer
Description: Markers of coagulation activation
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 18 | 18 | 16
percentage change from baseline | 12.6 [-3.3 to 28.4] | 2.4 [-14.0 to 18.7] | -1.6 [-3.6 to 0.4]

9. Secondary Outcome: F1+2
Description: Change in plasma concentrations of F1+2 a marker of coagulation activation
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 18 | 18 | 16
percentage change from baseline | 24.1 [4.2 to 43.9] | -5.5 [-19.4 to 8.4] | -8.5 [-20.4 to 3.5]

10. Secondary Outcome: Thrombin Generation, ETP Endogenous Thrombin Potential
Description: Change from baseline in thrombin generation, measured by thrombin generation assay-Calibrated automated thrombogram
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 18 | 18 | 16
percentage change from baseline | 63.9 [51.4 to 76.3] | 26.4 [14.5 to 38.2] | 7.1 [-3.2 to 17.4]

11. Other Pre Specified Outcome: Anti Mullerian Hormone (AMH)
Description: Change in Serum concentrations of anti-mullerian hormone reflecting ovarian reserve from baseline to nine weeks
Time Frame: baseline and 9 weeks
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
Number analyzed (Participants) | 19 | 20 | 17
ng/mL | -0.8 [-1.4 to -0.2] | -0.4 [-0.7 to 0.004] | 0.07 [-0.3 to 0.4]

ADVERSE EVENTS:
Time Frame: 9 weeks. During the study period.
Arm/Group | Synthetic Estrogen + Progestin | Natural Estrogen + Progestin | Progestin-Only
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-04-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT02352090/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT02352090/SAP_001.pdf